CLINICAL TRIAL: NCT03352622
Title: Pharmacogenomic in Colombian Patients With Rheumatoid Arthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Antioquia (Other)
Collaborators: Hospital Pablo Tobón Uribe (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: Pharmacogenomic
Record Dates: First submitted 2017-11-10; First posted 2017-11-24 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2017-06

CONDITIONS: Pharmacological Action
Keywords: PHARMACOGENOMICS; POLYMORPHISM

STUDY DESIGN:
Intervention Model Description: CASES AND CONTROLS
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CASES (Active Comparator): Patients with RA with methotrexate therapy and inhibitors of tumor necrosis factor alpha (TNFα) infliximab, etanercept, adalimumab; That present problems of effectiveness
  Interventions: Other: CASES
- CONTROLS (Active Comparator): Patients with RA with methotrexate therapy inhibitors of tumor necrosis factor alpha (TNFα) infliximab, etanercept, adalimumab; No problems of effectiveness
  Interventions: Other: CONTROLS

INTERVENTIONS:
Other: CASES — Patients with RA with methotrexate therapy and inhibitors of tumor necrosis factor alpha (TNFα) infliximab, etanercept, adalimumab; That present problems of effectiveness.
  Other Names: NO RESPONDERS
  Arms: CASES
Other: CONTROLS — Patients with RA with methotrexate therapy inhibitors of tumor necrosis factor alpha (TNFα) infliximab, etanercept, adalimumab; No problems of effectiveness
  Other Names: RESPONDERS
  Arms: CONTROLS

SUMMARY:
The pharmacogenomics of the Colombian population with rheumatoid arthritis (RA), understood as the individual response to drugs depending on the genome of each patient, can be an explanation for the problems of effectiveness and safety that appear during the pharmacotherapeutic treatment of RA.

Currently, there are limited studies on the pharmacogenomics of the Colombian population; Therefore, it is necessary to identify and classify the genetic polymorphisms characteristic of Colombian patients with RA, which influence the response of methotrexate, infliximab, etanercept, adalimumab and thus contribute to precision medicine and medical prescription according to the Specificity of the genome of each patient.

This project aims to determine the association of genetic polymorphisms with the response to inhibitors of tumor necrosis factor alpha (TNFα) and methotrexate. To do this, a prospective study of cases and controls will be performed in patients in 3 hospital of Colombia with pharmacotherapeutic treatment of methotrexate, infliximab, etanercept, adalimumab, in monotherapy or combination therapy.

As a result, it is expected to contribute to the performance of specific genetic tests for RA and the generation of a pharmacogenomic basis of the Colombian population with RA.

DETAILED DESCRIPTION:
Rheumatoid arthritis is an important public health problem; In recent years better health outcomes have been achieved with the incorporation of synthetic and biological disease modifying drugs. However, problems of variability in response are reported, leading to ineffectiveness and adverse reactions in 30-40% of patients. In this sense, Pharmacogenomics, through the study of genetic variants of proteins involved in the pharmacokinetics and pharmacodynamics of drugs, becomes a way to maximize the efficacy and safety of pharmacotherapy.

This work aims to give an overview of the pharmacogenomics of rheumatoid arthritis and the possibility of using genetic tools to support the pharmacotherapeutic decision in the clinical consultation, in order to improve the response to treatment of this disease.

The relevance of this study is to provide the possibility of applying the candidate genes selected for their biological importance, either in the kinetics or by their relation in the pharmacological action, in the identification of individuals at risk of adverse effects or With probability of being resistant to the treatment. Therefore, it is expected that the information generated will be able to be used in daily clinical practice, contributing to identify the best therapeutic option (greater effectiveness and safety) in patients with rheumatoid arthritis. In addition, it is expected that this type of information will contribute to optimize the costs of care in this disease, which is classified in Colombia as a high cost pathology, in which medicines can reach up to 86% of the total cost.

Overall, individuals respond differently to drug therapy and no medication is 100% effective in all patients, which may be due to an alteration in the pharmacokinetics and pharmacodynamics of drugs associated with conditions Genetic-environmental. In this context, the study of candidate pharmacogenomic genes has been most successful in identifying and explaining variation in pharmacological response, compared to candidate gene investigations of the disease. Therefore, this work should contribute to the choice of the best therapeutic option in patients with RA in Colombia and, thus, to strengthen the country's health sector.

ELIGIBILITY:
Inclusion Criteria:

* Patients with rheumatoid arthritis on treatment with Methotrexate, Adalimumab, Infliximab or Etanercept (monotherapy or combination therapy)
* Over 18 years
* With DAS 28 (Disease Activity Score in 28 Joints) greater than 3.2
* With SDAI (Simple Disease Activity Index) less than 3.3
* Use of medication> 3 months
* Anti TNFα, used for the first time.
* Subscribe to informed consent

Exclusion Criteria:

* Patients who after applying the tool to identify other causes of variability; Identify other causes that variability in response (non-adherence to travel, forgetfulness, etc.).
* Previous use of anti TNFα drugs.
* Inpatient Patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 372 (Estimated)
Dates: Start 2017-10-17 (Actual); Primary Completion 2018-10-17 (Estimated); Study Completion 2020-09-17 (Estimated)

PRIMARY OUTCOMES:
Number of exomes and genetic variants identified | 1 year
  The identification of polymorphisms will be carried out through the next generation sequencing technique

CONTACTS AND LOCATIONS:
Overall Officials: Yolima Puentes, Pharmacist, Principal Investigator — Universidad de Antioquia
Locations (1):
- Pablo Tobon Uribe Hospital, Medellín, Colombia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Salazar J, Moya P, Altes A, Diaz-Torne C, Casademont J, Cerda-Gabaroi D, Corominas H, Baiget M. Polymorphisms in genes involved in the mechanism of action of methotrexate: are they associated with outcome in rheumatoid arthritis patients? Pharmacogenomics. 2014 Jun;15(8):1079-90. doi: 10.2217/pgs.14.67. PMID 25084201
- [Background] Muralidharan N, Antony PT, Jain VK, Mariaselvam CM, Negi VS. Multidrug resistance 1 (MDR1) 3435C>T gene polymorphism influences the clinical phenotype and methotrexate-induced adverse events in South Indian Tamil rheumatoid arthritis. Eur J Clin Pharmacol. 2015 Aug;71(8):959-65. doi: 10.1007/s00228-015-1885-0. Epub 2015 Jun 14. PMID 26071279
- [Background] Dupont JA. Significance of operative cultures in total hip arthroplasty. Clin Orthop Relat Res. 1986 Oct;(211):122-7. PMID 3769251
- [Background] Bernzweig EP. Liability for malpractice...its role in nursing education. J Nurs Educ. 1969 Apr;8(2):33-41. No abstract available. PMID 4388501